CLINICAL TRIAL: NCT05750888
Title: Effects of Integrated Foot Core Strengthening With Exerciser Device on Balance Control and Walking in the Elderly With and Without Sarcopenia
Brief Title: Foot Core Exercise Program on Balance Control and Walking in Aged Sarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: P00001837
Record Dates: First submitted 2022-11-21; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2022-11

CONDITIONS: Sarcopenia; Muscle Weakness; Walking, Difficulty; Balance Control
Keywords: Foot core system; Intrinsic foot muscle; Balance control; 3D printing; Gait
MeSH Terms: conditions — Sarcopenia; Muscle Weakness; Mobility Limitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): A novel-designed intrinsic foot muscle-strengthening exerciser using 3D printing techniques will be used in the experimental group.
  Interventions: Behavioral: integrated exercise therapy with 3D printing exerciser for training intrinsic foot muscles
- Experimental group 2 (Sham Comparator): A regular exercise program will be provided in this group.
  Interventions: Behavioral: regular exercises for the elderly
- Control group (No Intervention): There is no exercise or other intervention in this group.

INTERVENTIONS:
Behavioral: integrated exercise therapy with 3D printing exerciser for training intrinsic foot muscles — The therapeutic exercise program with a custom-made 3-D printing foot core exerciser, consisting of warm-up exercise, active range of motion in the foot and ankle joints, foot core system strengthening program using the 3D printing device, and stretching exercises for foot and ankle.
  Other Names: novel foot core exercise program
  Arms: Experimental group 1
Behavioral: regular exercises for the elderly — The regular exercise provided for the elderly in the dwelling community, including walking, simple aerobic exercises, stretching exercises
  Other Names: regular exercises
  Arms: Experimental group 2

SUMMARY:
In modern society with an increasing aging population, recent literature has defined sarcopenia as a significant reduced mass and function of skeletal muscle with physical limitations due to aging. Clinically and experimentally, the foot often plays a crucial role in sensorimotor control and movement performance in standing, walking, and running. Apparently, previous literature has shown that the intrinsic and extrinsic foot muscles have significantly reduced muscle morphology and muscle strength in the elderly compared to that of young healthy controls. How to effectively increase foot muscles using muscle-strengthening exercises will be a crucial issue for further research and clinical intervention in this population.

The intrinsic foot muscles (IFM) are the primary local stabilizer to provide static and dynamic stability in the foot, which are part of the active and neural subsystems to constitute the foot core system. The intrinsic foot muscles (IFMs) may play a key role in supporting foot arches (e.g., the medial longitudinal arch, MLA), providing flexibility, stability, shock absorption to the foot, and partially controlling foot pronation. Due to the difficulties in teaching and learning the plantar intrinsic foot muscle (IFM) exercise, the accuracy and follow-up after learning this exercise could be questioned following this exercise program. Physiologically, the effects of integrated exercise intervention may be achieved following more than 4-week intensive exercise intervention at least. How to learn and activate this kind of exercise efficiently and effectively is a key issue for employing these exercise interventions in the elderly with and without sarcopenia.

In this project, we will aim to employ the novel intrinsic foot muscle strengthening device using 3-D printing techniques and to examine the feasibility and reliability of the morphology in intrinsic and extrinsic foot muscles and foot posture before and after exercise intervention using sonographic imaging and foot posture index in the elderly with and without sarcopenia; second, we will investigate whether the immediate and persistent increase in balance control and level-walking after this therapeutic exercise with novel 3-D printing foot core exerciser.

DETAILED DESCRIPTION:
In modern society with an increasing aging population, Asian Working Groups for Sarcopenia (AWSG) has defined sarcopenia as a significantly reduced mass and function of skeletal muscle with physical limitations due to aging. The prevalence in the globe has reported 5% - 25.7% of the elderly population and its associations are very high between daily activity limitations, physical limitations, and premature death. Clinically and experimentally, the foot often plays a crucial role in sensorimotor control and movement performance in standing, walking, and running. Apparently, previous literature has shown that the intrinsic and extrinsic foot muscles have significantly reduced muscle morphology and muscle strength in the elderly compared to that of young healthy controls. How to effectively increase foot muscles using muscle-strengthening exercises will be a crucial issue for further research and clinical intervention in this population.

Anatomically, the intrinsic foot muscles (IFM) are the primary local stabilizer to provide static and dynamic stability in the foot, which are part of the active and neural subsystems to constitute the foot core system. The intrinsic foot muscles (IFMs) may play a key role in supporting foot arches (e.g. the medial longitudinal arch, MLA), providing flexibility, stability, shock absorption to the foot, and partially controlling foot pronation. Due to the difficulties in teaching and learning the plantar intrinsic foot muscle (IFM) exercise, the accuracy and follow-up after learning this exercise could be questioned following this exercise program; Physiologically, the effects of integrated exercise intervention may be achieved following more than 4-week intensive exercise intervention at least. How to learn and activate this kind of exercise efficiently and effectively is a key issue for employing these exercise interventions in the elderly with and without sarcopenia.

This project consists of two main parts - first, we will aim to employ the novel intrinsic foot muscle strengthening device using 3-D printing techniques and to examine the feasibility and reliability of the morphology in intrinsic and extrinsic foot muscles and foot posture before and after exercise intervention using sonographic imaging and foot posture index in the elderly with and without sarcopenia; second, we will investigate whether the immediate and persistent increase in balance control and level-walking after this therapeutic exercise with novel 3-D printing foot core exerciser. More importantly, we elucidate important clinical evidence-based information of long-term novel therapeutic exercise intervention for clinicians and health policymakers.

ELIGIBILITY:
Inclusion Criteria:

* the elderly with sarcopenia [1, 2] Age is more than 65 years with a medical diagnosis of sarcopenia Be able to independently stand and walk To meet the criteria of the definition of sarcopenia in the AWGS 2019 consensus update on sarcopenia diagnosis and treatment Be able to understand independently the participation consent in this research project
* Healthy elder individuals A neutral foot alignment: determined by measurement of the resting calcaneal stance position (RCSP: between 2˚of inversion and 2˚of eversion) and scores on the navicular drop (ND: between 5 and 9 mm) test.

Foot Posture Index (FPI) Score is between 0 and 5. No pain in the lower limbs No history of lower limb injury that has affected function or caused the individual to seek previous medical or therapeutic intervention within 6 months

Exclusion Criteria:

* All groups not be able to sign the consent form for the participation Traumatic injury to lower limbs which impacted joint integrity and function (i.e., fractures) resulting in at least 1 interrupted day of desired physical activity Major neurological, cardiorespiratory, or circulatory disorders contribute to not being able to independently stand and walk.

Recent intervention/management within the last 6 months

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — The studies will involve individuals between 65-95 years of age with planned male to female ratio of 1:1
Enrollment: 60 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Sonographic imaging for cross-sectional area of muscles | changes among baseline, 4, 8 and 12 weeks
  The diagnostic ultrasound will be employed to detect the cross-sectional area (CSA) in specific foot intrinsic and extrinsic muscles, such as extrinsic muscle (Flexor digitorum longus FDL, Flexor Hallucis Longus FHL, and Peroneal longus PL) and intrinsic muscle ( Abductor Hallucis AbdH, Flexor Digitorum Brevis FDB and Flexor Hallucis Brevis FHB) CSA. The unit is cm2
Sonographic imaging for the width and thickness of muscles | changes among baseline, 4, 8 and 12 weeks
  The diagnostic ultrasound will be employed to detect the width and thickness of specific foot intrinsic and extrinsic muscles, such as extrinsic muscles (FDL, FHL, and PER) and intrinsic muscle (AbdH, FDB, and FHB)width and thickness, and plantar fascia thickness (at the heel, mid and forefoot sites). The unit is cm (the width and length)
Balance test for standing posture for area of sway trajectory in center of pressure (CoP) and center of mass (CoM) | changes among baseline, 4, 8 and 12 weeks
  A complete lower limb model will be established through commercial motion analysis software. Motion Analysis System with 12 optoelectronic cameras and two high-speed video cameras with two force plates will be used for further analysis in standing and level walking. Static postural control will be assessed in a quiet standing task on the two force plates to measure the variables of the center of pressure (CoP) and center of mass (CoM) at eyes-open and eyes-closed conditions. The unit is mm.
Balance test for standing posture for the velocity of sway trajectory in center of pressure (CoP) and center of mass (CoM) | changes among baseline, 4, 8 and 12 weeks
  A complete lower limb model will be established through commercial motion analysis software. Motion Analysis System with 12 optoelectronic cameras and two high-speed video cameras with two force plates will be used for further analysis in standing and level walking. Static postural control will be assessed in a quiet standing task on the two force plates to measure the variables of the center of pressure (CoP) and center of mass (CoM) at eyes-open and eyes-closed conditions. The unit is mm/sec.
Balance test for standing posture for the length of sway trajectory in center of pressure (CoP) | changes among baseline, 4, 8 and 12 weeks
  A complete lower limb model will be established through commercial motion analysis software. Motion Analysis System with 12 optoelectronic cameras and two high-speed video cameras with two force plates will be used for further analysis in standing and level walking. Static postural control will be assessed in a quiet standing task on the two force plates to measure the variables of the center of pressure (CoP) and center of mass (CoM) at eyes-open and eyes-closed conditions. The unit is mm.
Functional walking test for spatio-temporal parameters | changes among baseline, 4, 8 and 12 weeks
  Spatio-temporal parameters will be calculated during level walking. The subject will be asked to walk at slow, self-paced, and fast walking using a metronome. The unit is m/sec.
Functional walking test for joint kinematics in the lower limb | changes among baseline, 4, 8 and 12 weeks
  Joint kinematic data will be calculated during level walking. The subject will be asked to walk at slow, self-paced, and fast walking using a metronome. The unit is degree.
Functional walking test for joint kinetics in the lower limb | changes among baseline, 4, 8 and 12 weeks
  Joint kinetic data will be calculated during level walking. The subject will be asked to walk at slow, self-paced, and fast walking using a metronome. The unit is Nm.
Clinical Questionnaires for assessment in physical capacity in the elderly | changes among baseline, 4, 8 and 12 weeks
  Short Physical Performance Battery (0-12) questionnaires will be employed in this study. The unit is a unit on a scale.
Clinical Questionnaires for assessment in functional capacity and falling condition in the elderly | changes among baseline, 4, 8 and 12 weeks
  Strength, Assisting with walking, Rising from a chair, Climbing stairs, and Falling questionnaire (0-10) will be employed in this study. The unit is a unit on a scale.
Clinical Questionnaires for assessment in functional capacity and strength condition in the elderly | changes among baseline, 4, 8 and 12 weeks
  Strength, Assisting with walking, Rising from a chair, Climbing stairs, and Calf circumference (0-20). The unit is a unit on a scale.

SECONDARY OUTCOMES:
Clinical Questionnaires for assessment in cognitive capacity in the elderly | changes among baseline, 4, 8 and 12 weeks
  Mini-Mental State Examination (0-30) questionnaires will be employed in this study. The unit is a unit on a scale.
Clinical Questionnaires for assessment in nutritional status in the elderly | changes among baseline, 4, 8 and 12 weeks
  Mini Nutritional Assessment - Short Form (0-11) will be employed in this study. The unit is a unit on a scale.
Clinical Questionnaires for assessment in frail status in the elderly | changes among baseline, 4, 8 and 12 weeks
  Frail Index (0.0-1.0) will be employed in this study. The unit is a unit on a scale.
Clinical Questionnaires for assessment in frailty condition the elderly | changes among baseline, 4, 8 and 12 weeks
  A clinical Frailty Scale (1-9) will be employed in this study. The unit is a unit on a scale.

CONTACTS AND LOCATIONS:
Overall Officials: Chich-Haung R Yang, PhD, Principal Investigator — College of Medicine, Tzu Chi University
Locations (1):
- BuddhistTCGH, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Dufour AB, Hannan MT, Murabito JM, Kiel DP, McLean RR. Sarcopenia definitions considering body size and fat mass are associated with mobility limitations: the Framingham Study. J Gerontol A Biol Sci Med Sci. 2013 Feb;68(2):168-74. doi: 10.1093/gerona/gls109. Epub 2012 Apr 13. PMID 22503991
- [Derived] Kao SL, Hsiao ML, Wang JH, Chen CS, Chen SY, Shiau YJ, Yang CH. Effects of integrated intrinsic foot muscle exercise with foot core training device on balance and body composition among community-dwelling adults aged 60 and above. BMC Geriatr. 2024 May 7;24(1):403. doi: 10.1186/s12877-024-04945-y. PMID 38714957